CLINICAL TRIAL: NCT04690972
Title: "Constitution of a Biological Collection to Establish Preclinical Translational Models for the Study of Tumors and Chronic Liver Diseases".
Acronym: LivMOD
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-76
Record Dates: First submitted 2020-12-04; First posted 2020-12-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Liver Disease and Cirrhosis; Liver Cancer; Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Viral Hepatitis B; Viral Hepatitis C; Viral Hepatitis D
Keywords: Liver disease; Ex vivo models; Single cell; Biomarkers; Spheroïds
MeSH Terms: conditions — Fibrosis; Liver Neoplasms; Non-alcoholic Fatty Liver Disease; Hepatitis B; Hepatitis C; Hepatitis D; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample Cohort 1 and 2 : 1 tube (10ml) of blood Cohort 3 : 10 tubes (10ml) of blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hepato-bilio-pancreatic surgery: Patients whom hepato-bilio-pancreatic surgery is indicated as part of the care
  Interventions: Procedure: Blood sample during surgery
- biopsy of the hepatic parenchyma: Patients whom a biopsy of the hepatic parenchyma, one or more hepatic nodules or a loco-regional treatment is indicated as part of the care
  Interventions: Procedure: Taking an additional biopsy
- Viral chronic infection: Patients with a viral chronic liver disease
  Interventions: Diagnostic Test: Blood sample during diagnostic test

INTERVENTIONS:
Procedure: Blood sample during surgery — During the hepato-bilio-pancreatic surgery, blood is drawn.
  Groups: Hepato-bilio-pancreatic surgery
Procedure: Taking an additional biopsy — As part of the treatment, an additional biopsy is executed and blood is drawn.
  Other Names: Blood sample during biopsy
  Groups: biopsy of the hepatic parenchyma
Diagnostic Test: Blood sample during diagnostic test — Blood sample as part of the care
  Groups: Viral chronic infection

SUMMARY:
Development of preclinical translational models for chronic liver tumors and diseases study, such as spheroids cultured in autologous medium and murine xenograft models to test the efficacy of new therapeutic strategies.

DETAILED DESCRIPTION:
The Institute for Research on Viral and Hepatic Diseases, Inserm Unit UMR_S 1110, in Strasbourg, studies hepatic diseases such as non-alcoholic steatohepatitis (NASH), non-alcoholic fatty liver disease (NAFLD), cirrhosis and hepatocellular carcinoma (CHC). These diseases can be induced by hepatitis viruses, B (HBV), C (HCV) and D (VHD), but also a poor lifestyle combining overeating and the sedentary lifestyle of our current living patterns.

To date, no treatment is available to cure non-alcoholic steatohepatitis (NASH), cirrhosis, and prevent the development of liver tumors. One of the reasons for the lack of specific treatment is the limited knowledge of the pathophysiology of the liver and the hepatic microenvironment. In addition, the heterogeneity of HCC and associated underlying liver diseases, and the lack of adequate preclinical models are at the root of the difficulties in identifying an effective therapeutic target for these diseases.

Thus, new molecular profiling techniques and strategies are needed to meet these medical needs, in particular the prediction of the response to treatment of HCC, which is still largely unsatisfactory, and the discovery of new therapeutic targets. Using innovative approaches, UMR_S 1110 utilizes single cell RNA sequencing, which is a high resolution technique to analyze gene expression at the individual cell level. This technique represents the most advanced tool for studying heterogeneous tissues such as cancerous tissue.

An in-depth knowledge of HCC and the liver tumor environment at the single-cell level is crucial for understanding the progression of liver disease, for identifying new therapeutic targets and improving clinical outcomes by allowing for estimate the response to treatment and thus improve the patient's vital prognosis, by offering him an adapted personalized treatment. In order to identify factors determining hepatocarcinogenesis, predictors of response to treatment and new therapeutic targets, the investigators propose to analyze tissues from patients with chronic liver disease.

The investigator aim :

1. / to establish ex vivo models of chronic hepatic disease and hepatic tumors, in order to study and validate the therapeutic targets identified in the laboratory from single cell RNA sequencing from hepatic tissues obtained from patients. These models include spheroid cultures and models of mice developing liver tumors from xenografts of tumors from patients. To ensure the successful establishment of these complex models, the use of autologous sera is necessary.
2. / profile the hepatic tumors and the hepatic tissue adjacent to the tumor, the site of chronic liver disease, using single-cell RNA sequencing in order to study the heterogeneity and complexity of the tumor, to identify novel therapeutic targets and tumor phenotypes that correlate with response to treatment.

Patient-derived preclinical models, developed at unit UMR_S1110, will allow us to better understand the biology of chronic liver disease and liver tumors at the patient level, identify the most appropriate treatment for the patient, and evaluate new treatments and biomarkers to non-invasively diagnose the onset of liver disease, for the benefit of personalized medicine for the benefit of the patient.

Blood samples obtained from patients with chronic liver disease will also allow us to:

* Advance knowledge on viral hepatitis, in particular HCV, HBV and HDV;
* Implement new strategies for the development of a vaccine for HCV;
* Identify new biomarkers of hepatic carcinogenesis by comparing the metabolomic and inflammatory profiles of patients.

The partnership between Inserm, the University of Strasbourg and the University Hospitals of Strasbourg makes it possible to create unique synergies that will ultimately help identify new targets for therapeutic and preventive strategies against these diseases which represent a major public health problem.

ELIGIBILITY:
Inclusion Criteria:

1. Patients

   * diagnosed with chronic liver disease (viral or not)
   * diagnosed with at least one liver nodule for which a biopsy is planned as part of the care
   * for hepatobiliary surgery planned as part of care
   * for locoregional treatment for HCC is indicated
2. Patients able to receive and understand information relating to the study and give their written informed consent
3. Patients affiliated to the French social security system

Exclusion Criteria:

1. Minor patients
2. Patients under legal protection,
3. Patients subject to legal protection or unable to express their consent,
4. Patients in a situation of social fragility,
5. Pregnant or breastfeeding woman,
6. No signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with hepato-bilio-pancratic disease (tumor, viral infection, injury)
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
Surgery for a hepato-bilio-pancreatic issue | through study completion, an average of 8 year
  Patients whom hepato-bilio-pancreatic disease

CONTACTS AND LOCATIONS:
Locations (1):
- PU-PH, Directeur de l'UMR_S1110 Unité Inserm d'affiliation : UMR_S1110, Strasbourg, France